CLINICAL TRIAL: NCT05736510
Title: The Effect of Binaural Sound on Recovery of General Anesthesia in Patients Undergoing Laparoscopic Simple Gynecological Surgery
Brief Title: Brainwave Entrainment During Emergence
Acronym: BB_emergence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2212-028-1383
Record Dates: First submitted 2023-02-02; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, General
Keywords: Brain Waves; anesthesia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A prospective randomized study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binaural (Experimental): Exposed to binaural sound (40 Hz) from the end of pneumoperitoneum until the eyes are open
  Interventions: Other: Binaural sound
- Control (Active Comparator): Applied silent files from the end of pneumoperitoneum until the eyes are open
  Interventions: Other: Control

INTERVENTIONS:
Other: Binaural sound — When the pneumoperitoneum ends, the anesthesiologist puts headphones on the patient and plays the allocated file. In the experimental group, the allocated file is binaural sound with 40Hz beat. Thereafter, the target of PSI is to be between 40 and 50. If the Psi increases above 50, increase the propofol concentration by 0.5 mg/mL and record it. Train of four counts keep between 1 to 3 (moderate block). When the operation is ended, stop anesthetics administration, and, we reverse neuromuscular blocking using sugammadex (2mg/ kg). When the anesthesiologist starts waking the patient up, call the patient's name (unify into "OOO, open your eyes."). The anesthesiologist lightly tap the patient's shoulder and avoid excessive sound or stimulation.
  Arms: Binaural
Other: Control — When the pneumoperitoneum ends, the anesthesiologist puts headphones on the patient and plays the allocated file. In the control group, the allocated file is silent. Thereafter, the target of PSI is to be between 40 and 50. If the Psi increases above 50, increase the propofol concentration by 0.5 mg/mL and record it. Train of four counts keep between 1 to 3 (moderate block). When the operation is ended, stop anesthetics administration, and, we reverse neuromuscular blocking using sugammadex (2mg/ kg). When the anesthesiologist starts waking the patient up, call the patient's name (unify into "OOO, open your eyes."). The anesthesiologist lightly tap the patient's shoulder and avoid excessive sound or stimulation.
  Arms: Control

SUMMARY:
The investigators will compare whether there is a significant difference in the time required for general anesthesia recovery according to application of the binaural sound after surgery.

DETAILED DESCRIPTION:
After entering the operating room, electrocardiogram, pulse oxygen saturation, blood pressure meter, and sedline are attached to start monitoring vital signs and patient state index (PSI). propofol and the remifentanil continuous infusion device is connected as close as possible to the catheter insertion site. Anesthesia is induced with total intravenous anesthesia (4 ng/mL of Remifentanil, 4 mg/mL of propofol). Rocuronium is administered after checking the patient's unconsciousness. When appropriate neuromuscular blocking is reached, tracheal intubation is performed. The anesthesia maintenance is performed to keep stable vital sign and PSI between 25 and 50. End-tidal carbon dioxide is controlled to be between 30 mmHg and 40 mmHg.

When the pneumoperitoneum ends, the propofol concentration is recorded (T0). The anesthesiologist in charge of anesthesia puts headphones on the patient and plays the allocated file. The allocated file is named the screening number. Depending on the allocated group, the audio file is binaural sound for the experimental group, and a silent file for the control group.

The anesthesiologist cannot know group allocation, since the length and size of files are the same. Thereafter, the target of PSI is to be between 40 and 50. If the Psi increases above 50, increase the propofol concentration by 0.5 mg/mL and record it. Train of four counts keep between 1 to 3 (moderate block). When the operation is ended, stop anesthetics administration, and record the time (T1). At the same time, the investigators reverse neuromuscular blocking using sugammadex (2mg/ kg).

When the anesthesiologist starts waking the patient up, call the patient's name (unify into "OOO, open your eyes."). The anesthesiologist lightly tap the patient's shoulder and avoid excessive sound or stimulation.

Record the time (T2) when the PSI reaches 50, the time when the patient opens eyes (T3), and the time (T4) when the extubation of endotracheal tube was done. T3-T1 is the time it took the patient to open his eyes (primary end point). Write the effect site concentration of propofol and remifentanil recorded for each time points.

The patient's sedline EEG data from the end of pneumoperitoneum until the patient's exit operating room is collected as raw data. The patient's blood pressure and heart rate are measured at each time points. The investigators evaluate sedation and agitation of the patients using Ramsay Sedation Scale.

In the post-anesthesia care unit, pain score (NRS 0-10), postoperative nausea vomiting, medication, and length of stay are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 19 and 50 years of age who are scheduled to undergo laparoscopic salpingo-oophorectomy/ ovarian cystectomy
* Intellectual level to understand the procedures of the clinical trial
* Physical status classification of the American Society of Anesthesiology (ASA) 1-2 grades

Exclusion Criteria:

* Patients with hearing loss or using hearing aids
* Patients who have been given narcotic painkillers or sedative drugs within a week.
* Alcohol-dependent or drug-dependent patients
* Patients with drug hypersensitivity to anesthetics
* Patients with arrhythmia, cardiovascular disease, impaired heart function, decreased circulatory blood flow
* Patients with liver failure
* Patients with other major medical or psychological disorder that will affect the treatment response
* Patients with claustrophobia or anxiety disorder
* Patients with organic brain disorders or other conditions that cannot be properly measured by PSI
* Patients who have been newly diagnosed with myocardial infarction, cerebral ischemic seizure, stroke, clinically significant coronary artery disease, or have undergone percutaneous carotid coronary dilatation or coronary bypass treatment within 6 months
* Patients with a history of epilepsy or seizures
* Patients with acute angle glaucoma
* Patients who deemed unsuitable for this clinical trial

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Eye opening time | after the anesthetic infusion is terminated until 1 hour
  The time it takes to open patient's eyes in response to the voice after the anesthetic infusion is terminated.

SECONDARY OUTCOMES:
Extubation time | after the anesthetic infusion is terminated until 1 hour
  The time it takes from the end of the anesthetic infusion to the extubation of endotracheal tube
Systolic blood pressure | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  Noninvasive systolic blood pressure
Diastolic blood pressure | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  Noninvasive diastolic blood pressure
Mean blood pressure | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  Noninvasive mean blood pressure
Heart rate | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  Heart rate
alpha band activity | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  alpha band activity of electroencephalogram from Sedline data
beta band activity | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  beta band activity of electroencephalogram from Sedline data
theta band activity | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  theta band activity of electroencephalogram from Sedline data
delta band activity | from the end of the anesthetic infusion to the exit of operating room until 1 hour
  delta band activity of electroencephalogram from Sedline data
Ramsay Sedation Scale | When the end of anesthesia within 5minutes
  The degree of patient's sedation or agitation (1 to 6: 1 means "Patient is anxious and agitated or restless, or both"; 6 means "Patient exhibits no response")
Postoperative recovery score | When the patient stay in post-anesthesia care unit up to 1 hour
  Postoperative recovery score (0-10; activity (0-2), respiration (0-2), circulation (0-2), consciousness level (0-2), and color (0-2); optimum score 10)
Pain score | When the patient stay in post-anesthesia care unit up to 1 hour
  Postoperative pain score using numeric rating scale(0-10: 0, no pain; 10, worst possible pain)
Rate of postoperative nausea and vomiting | When the patient stay in post-anesthesia care unit up to 1 hour
  Rate of postoperative nausea and vomiting
Length of stay in post-anesthesia care unit | From entering to exit the post-anesthesia care unit up to 2 hours
  Length of stay in post-anesthesia care unit
Medication | When the patient stay in post-anesthesia care unit up to 1 hour
  Rate of administration of any medication in post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, MD.,PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid W, Marhofer P, Opfermann P, Zadrazil M, Kimberger O, Triffterer L, Marhofer D, Klug W. Brainwave entrainment to minimise sedative drug doses in paediatric surgery: a randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):330-335. doi: 10.1016/j.bja.2020.05.050. Epub 2020 Jul 8. PMID 32653082
- [Background] Ozkose Z, Yalcin Cok O, Tuncer B, Tufekcioglu S, Yardim S. Comparison of hemodynamics, recovery profile, and early postoperative pain control and costs of remifentanil versus alfentanil-based total intravenous anesthesia (TIVA). J Clin Anesth. 2002 May;14(3):161-8. doi: 10.1016/s0952-8180(01)00368-3. PMID 12031745